CLINICAL TRIAL: NCT01395394
Title: The Ability of Kuvan® (Sapropterin Dihydrochloride) to Prevent Meal-induced Lipid Peroxidation and Endothelial Dysfunction in Patients With Phenylketonuria: a Pilot Study
Brief Title: Phenylketonuria, Oxidative Stress, and BH4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with recruitment and agreed with Sponsor to report completed data as case reports
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Rani Singh, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB00046153
Record Dates: First submitted 2011-06-23; First posted 2011-07-15 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; PKU; tetrahydrobiopterin; sapropterin dihydrochloride; BH4; Kuvan; Oxidative stress
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BH4 Non-Responders (Experimental): Participants in this group have PKU and were deemed unresponsive to the drug. They will attend their first study visit, and proceed through the meal challenge without BH4. They will then take BH4 for 2 weeks. The second meal challenge will be performed with the participant's final dose of BH4.
  Interventions: Drug: Kuvan; Other: Meal Challenge
- Healthy Controls (Experimental): Participants in this group match an enrolled PKU participant in terms of age, gender, and body mass index class. They will participate in a single study visit and will not be given BH4.
  Interventions: Other: Meal Challenge
- BH4 Responders (Experimental): Participants in this group will use their already prescribed BH4 with the meal challenge and be assessed at a single study visit. They will take their prescribed BH4 with the meal.
  Interventions: Other: Meal Challenge

INTERVENTIONS:
Drug: Kuvan — Participants in the BH4 Non-Responder group will be given a 20 mg/kg body weight/day dose of Kuvan to take on a daily basis for two weeks. The last dose will be administered at the participant's study visit 2.
  Other Names: Sapropterin dihydrochloride; tetrahydrobiopterin; BH4
  Arms: BH4 Non-Responders
Other: Meal Challenge — At each study visit, patients will receive a meal high in polyunsaturated fats that will promote a transitory increase in oxidative stress measures and endothelial dysfunction

SUMMARY:
The purpose of this study is to see how tetrahydrobiopterin therapy (BH4; also known as sapropterin dihydrochloride or Kuvan) affects measures of oxidative stress and endothelial function in patients with Phenylketonuria (PKU).

DETAILED DESCRIPTION:
Oxidative stress will be induced by having participants eat a meal in polyunsaturated fats. The investigators will see how participants respond to the meal challenge over the course of 6 hours.

* PKU participants who are currently on BH4 therapy will be evaluated while taking BH4 with the meal at a single study visit.
* PKU participants who did not responded to BH4 therapy will be evaluated twice. At the first study visit the investigators will see how you react to the meal challenge when you are not given BH4. You will be given BH4 for two weeks, then return for a second meal challenge study visit while taking BH4.
* Healthy controls will be evaluated after consuming the meal only (no BH4) at a single study visit.

ELIGIBILITY:
Inclusion Criteria:

* Have read, understood, and signed this consent form (and assent form, if <18 years old)
* Are between the ages of 10-45 years
* Weigh at least 75 pounds (34 kg)
* Meet group-specific criteria

Exclusion Criteria:

* Smoke
* Have any history of cardiovascular disease
* Have hepatic impairment, or demonstrate abnormal baseline liver function lab test results
* Have donated blood within 3 months prior to the study or are anemic as shown by the baseline lab results
* Are unwilling to discontinue dietary supplements (excluding medical food) two weeks prior to their first study visit
* Are currently take medications that will interfere with the interpretation of selected endpoints (such as lipid-lowering medication)
* Are currently pregnant or breastfeeding
* Excluding PKU, have a chronic illness, disorder, or condition (including but not limited to diabetes, hypertension, cancer)
* Have taken any investigational drug (including Kuvan for Kuvan-unresponsive participants & controls) within 3 months prior to the study
* In the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rani H Singh, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Decatur, Georgia, United States

REFERENCES:
- See also: Study Website — http://www.genetics.emory.edu/nutrition/pbos

RESULTS

PARTICIPANT FLOW:
Period: Baseline Study Visit
Arm/Group | BH4 Non-Responders | Healthy Controls | BH4 Responders
Started | 4 | 3 | 5
Completed | 3 | 3 | 5
Not Completed | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Study Visit 2 (Non-responders Only)
Arm/Group | BH4 Non-Responders | Healthy Controls | BH4 Responders
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BH4 Non-Responders | Healthy Controls | BH4 Responders | Total
Number analyzed (Participants) | 4 | 3 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (13.4) | 33.5 (15.7) | 18.5 (3.8) | 27.4 (12.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2 | 4
  Between 18 and 65 years | 3 | 2 | 3 | 8
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 3 | 2 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 5 | 12
high-sensitivity CRP [Mean (Standard Deviation); unit: mg/L] | 1.3 (1.2) | 0.61 (0.14) | 1.04 (1.48) | 1.06 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: Lipid Peroxidation
Description: Markers will be assessed every other hour for each 6-hour study visit. Kuvan responders and healthy controls will only be assessed at one 6-hour study visit. Kuvan non-responders will be assessed at two study visits (a baseline visit, and a visit after two weeks of Kuvan therapy). Values will be assessed groupwise and also assessed for intrapersonal change in the Kuvan non-responsive group. Time frame of participation is estimated at one month.
Time Frame: Lipid peroxidation will be measured every other hour for six hours at baseline (study visit 1) for all study groups
Population: Study was terminated due to difficulty recruiting patients, thus analysis was limited to preliminary data on 11 patients only. TBARS was measured in 3 BH4 responders only - data were unavailable for 8 other participants (2 responders, 3 non-responders, and 3 controls) due to inadequate sample volume.
Measure: Mean (Standard Deviation); unit: umole/L
Arm/Group | BH4 Non-Responders | Healthy Controls | BH4 Responders
Number analyzed (Participants) | 0 | 0 | 3
umole/L
  Baseline (prior to meal challenge) |  |  | 0.57 (0.33)
  2-hours post meal |  |  | 0.62 (0.53)
  4-hours post meal |  |  | 0.73 (0.39)
  6-hours post meal |  |  | 0.78 (0.47)

2. Primary Outcome: C-Reactive Protein (CRP)
Description: as for outcome 1
Time Frame: CRP will be measured every other hour for six hours at baseline (study visit 1) for all study groups and again during a second visit 2 weeks after baseline in BH4 Non-Responders only (study visit 2)
Population: Study was terminated due to difficulty recruiting patients, thus analysis was limited to preliminary data on 11 patients only. CRP was measured in 10 subjects - data were unavailable for 1 control participant due to inadequate sample volume.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | BH4 Non-Responders | Healthy Controls | BH4 Responders
Number analyzed (Participants) | 3 | 2 | 5
mg/dl
  Baseline, prior to meal challenge (n=3, 2, 5) | 1.46 (1.47) | 0.61 (0.14) | 1.04 (1.48)
  2-hours post meal (n=3, 2, 5) | 1.50 (1.49) | 0.58 (0.12) | 0.99 (1.40)
  4-hours post meal (n=3, 2, 5) | 1.55 (1.50) | 0.55 (0.18) | 0.96 (1.33)
  6-hours post meal (n=3, 2, 5) | 1.59 (1.60) | 0.55 (0.11) | 0.90 (1.24)
  Baseline V2, prior to meal challenge (n=3, 0, 0) | 1.51 (1.56) | NA (NA) — Controls did not complete Study Visit 2 | NA (NA) — BH4 Responders did not complete Study Visit 2
  2-hours post meal (V2; n=3, 0, 0) | 1.55 (1.67) | NA (NA) — Controls did not complete Study Visit 2 | NA (NA) — BH4 Responders did not complete Study Visit 2
  4-hours post meal (V2; n=3, 0, 0) | 1.79 (2.11) | NA (NA) — Controls did not complete Study Visit 2 | NA (NA) — BH4 Responders did not complete Study Visit 2
  6-hours post meal (V2; n=3, 0, 0) | 1.58 (1.69) | NA (NA) — Controls did not complete Study Visit 2 | NA (NA) — BH4 Responders did not complete Study Visit 2

ADVERSE EVENTS:
Arm/Group | BH4 Non-Responders | Healthy Controls | BH4 Responders
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/5

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No